CLINICAL TRIAL: NCT01359059
Title: Pre- vs. Post-incisional Pregabalin for Postoperative Pain Attenuation and Analgesics Spare in Orthopedic Oncologic Patients: A Comparative, Randomized, Double Blind Study Protocol
Brief Title: Pre- Versus Post-incisional Pregabalin for Postoperative Pain Attenuation and Analgesics Spare in Orthopedic Oncologic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Avi A Weinbroum, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TASMC-11-HF-0248-11-CTIL
Record Dates: First submitted 2011-05-18; First posted 2011-05-24 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Postoperative Pain
Keywords: assess the beneficial effects of PGL administered either pre or post surgery; assess the satisfaction rate in the orthopedic oncologic patients
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- IV-PCA (Patient-controlled analgesia) morphine (Active Comparator)
  Interventions: Drug: Pregabalin
- Patient controlled epidural analgesia (PCEA) fentanyl (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Patients in one set (40 patients/set) will receive 150 mg of PGL or placebo at 20:00 the evening before surgery and 1.5 h before surgery and will undergo surgery under GA. The 2nd set of patients will be randomized similarly but will undergo surgery under epidural analgesia. One physician whose duty in the study will end at the point of preoperative preparation will provide the patients with the preemptive drug. No other premedication will be administered to any patient. Post-operatively, patients who received preoperative PGL patients will be given placebo while the pre-surgery-placebo-treated ones will receive PGL, all at 2 h after surgery. All patients will then be given 150 mg twice daily thereafter, Q 12 h postoperatively up to 96 h.
  Arms: IV-PCA (Patient-controlled analgesia) morphine
Drug: Pregabalin — Patients in one set (40 patients/set) will receive 150 mg of PGL or placebo at 20:00 the evening before surgery and 1.5 h before surgery and will undergo surgery under GA. The 2nd set of patients will be randomized similarly but will undergo surgery under epidural analgesia. One physician whose duty in the study will end at the point of preoperative preparation will provide the patients with the preemptive drug. No other premedication will be administered to any patient. Post-operatively, patients who received preoperative PGL patients will be given placebo while the pre-surgery-placebo-treated ones will receive PGL, all at 2 h after surgery. All patients will then be given 150 mg twice daily thereafter, Q 12 h postoperatively up to 96 h.
  Arms: Patient controlled epidural analgesia (PCEA) fentanyl

SUMMARY:
Hypothesis

No studies considered the comparison of preemptive vs. post-surgery Pregabalin (PGL) only administration. The investigators believe that the administration of PGL preemptively would diminish pain sensation and therefore the need for opioids administration in orthopedic-oncologic patients more effectively than if administered starting postoperatively.

DETAILED DESCRIPTION:
Background

Proper pain relief is a major concern of patients worldwide. Pain concerns the surgical team as well, because of its correlation with clinical outcomes and patients' satisfaction rate. Studies have shown that negative clinical outcome with regard to pain control includes decreases in vital capacity and alveolar ventilation, pneumonia, tachycardia, hypertension, myocardial ischemia, transition into chronic pain, poor wound healing, and psychological sequelae. Pain has been found to be one of the three most common medical causes of delayed/aborted discharge after ambulatory surgery, the other two being drowsiness and postoperative nausea/vomiting. Despite progress that has been made with regard to postoperative pain control, and the development of new standards for pain control, many patients continue to experience intense pain after surgery.

Recent advances in the understanding of the particularities of central sensitization indicate that it plays an important role in post surgical and post traumatic pain and therefore should be avoided. We now distinguish postoperative pain, which is mostly nociceptive, and which perceives pain following surgical insult, from the exacerbation of acute nociceptive pain that leads to neural sensitization, when sensations that are not normally painful, are perceived as painful, as in hyperalgesia and allodynia. Thus, acute pain may transform into subacute or chronic pain, conditions that are harder to control when more persistent (chronic) they become. Better pain control, possibly using drugs that affect both acute and chronic pains, seems therefore the current optimal choice.

Multimodal analgesia Advances in knowledge of the neuropharmacological molecular mechanisms of pain have led to the development of "multimodal analgesia" practice.

The concept of multimodal analgesia is now a well established clinical practice. For example, non-steroidal anti-inflammatory medications combined with intravenous patient-controlled morphine administration, may decrease nausea and sedation in patients when compared with that using patient-controlled morphine analgesia alone. Multimodal analgesia also can produce opioid sparing effects. Our group has shown repeatedly, that multimodal analgesia spares postoperative morphine consumption and increases level of patients' satisfaction. However, they may not improve postoperative outcome in terms of faster recovery, reduced hospital stay, and decreased length of convalescence.

Analgesic adjuvant Adjuvants are compounds, which by themselves may have undesirable side effects or low potency but in combination with opioids allow a reduction of narcotic dosing for postoperative pain control. They are needed due to side effects of opioid analgesics, which hinder recovery, especially when increasingly utilizing ambulatory surgical procedures. One of the newer groups of products that are non-analgesic substances, therefore named "adjuvants", are anticonvulsants (e.g., pregabalin).

Pregabalin (PGL) Interest has been focused on the analgesic, sedative, anxiolytic, and opioid-sparing effects of pregabalin (PGL) (S+ 3-isobutyl GABA), a structural analog of GABA (Gamma-Aminobutyric Acid) and a derivative of gabapentin in various pain settings, including postoperative pain. Of a similar mechanism of action, it is thought to possess a superior pharmacokinetic profile than gabapentin. Pregabalin has a variable role in neuropathic pain conditions, such as post-herpetic neuralgia, painful diabetic neuropathy, central neuropathic pain, and fibromyalgia. Some studies had not demonstrated a significant analgesic effect in the acute, postoperative pain; others propose PGL to have effective sedative and opioid-sparing effects , both useful characteristics for the control of acute pain. Opioid sparing effects and improved pain scores have been seen after abdominal and pelvic surgery. Its many potential actions such as reducing opioid requirements, prevention and reduction of opioid tolerance, improvement of the quality of opioid analgesia, decreased respiratory depression, relief of anxiety, and gastric sparing, make it an attractive drug to consider for control of pain in the post operative period.

Population characteristics The orthopedic oncological patients are a specific group of individuals whose demand for antinociception starts rather before surgery because of the bone tumor-generated pain that usually signals the first existence of pathology. Subsequently, these patients would require postoperatively more analgesics than after general surgery and for a longer period of time. We have demonstrated previously that acute pain that is superimposed on an already aroused CNS (central nervous system), i.e., the presence of central sensitization, would create a situation where complete antinociception is hard to obtain, as in these patients, and therefore the efficacy of the antinociceptive protocol is best tested, comprised the possible transformation of acute into chronic pain.

preemptive drug has been pointed out as a beneficial tool for reducing perioperative pain. Various techniques have been employed for this purpose; different drugs were used as well. The beneficial effects of preemptive PGL were documented in patients who had undergone lumbar discectomy, both immediately and 1 and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients who will undergo bone with or without soft tissue cancer surgery type II and III [24,25] under general or epidural anesthesia in Tel-aviv Sourasky Medical Center will be enrolled to this study that will be approved by our institutional human research and ethics committee.
* All participants will sign a Helsinki-approved informed consent, and will be given full explanation of the drug, PCA and the numerical rating scale (NRS) during the pre-anesthesia interview.

Exclusion Criteria:

* These will include allergy to opioids, bupivacaine, midazolam, PGL, or non-steroidal anti-inflammatory drugs (NSAIDs), a history of chronic pain or psychiatric disorders and the use of centrally acting drugs of any sort. Patients <18 or >80 years, soldiers and pregnant women will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
To assess the beneficial effects of PGL administered either pre-incisionally or post-incisionally on the immediate and late (1- and 3 months) postoperative analgesia requirements and pain scores | 2 years
  In the PACU (post-anesthesia care unit), the parameters (pain, sedation, feeling of anxiety, total morphine, fentanyl, and bupivacaine consumptions, PCA activation, antinociceptives PO/IV, overall maximal pain intensity throughout the study period) will be assessed by the attending physician every 15 min for the first postoperative hour and every 30 min thereafter.
  On the ward, vital signs will be recorded Q 8 h.

CONTACTS AND LOCATIONS:
Overall Officials: Avi Weinbroum, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Weizman 6, Israel